CLINICAL TRIAL: NCT00191100
Title: Phase 3 Randomized Comparison of Concurrent Gemcitabine, Cisplatin, and Radiation Followed by Adjuvant Gemcitabine and Cisplatin Versus Concurrent Cisplatin and Radiation in Cancer of the Cervix Stages IIB to IVA
Brief Title: Comparative Study of Gemcitabine,Cisplatin and Radiation Versus Cisplatin and Radiation in Cancer of the Cervix
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4015; B9E-MC-JHQS
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-05-25 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Cancer of Cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Gemcitabine; Cisplatin; Brachytherapy

ARMS (2):
- 1 (Experimental): Cisplatin, 40 mg/m2, once weekly (QW), intravenous (IV), 6 weeks and Gemcitabine 125 mg/m2, once weekly (QW), intravenous (IV), 6 weeks and Pelvic radiation, 1.8 Gy/day, 5 days/week, 6 weeks
  Brachytherapy, 30-35 Gy over 1 week
  Two week rest period with no chemotherapy or radiation
  Cisplatin, 50 mg/m2, intravenous (IV), day 1 of 21 day cycle for two 21-day cycles and Gemcitabine, 1000 mg/m2, day 1 and day 8 for two 21 day cycles
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Radiation: Brachytherapy; Radiation: Pelvic radiation
- 2 (Active Comparator): Cisplatin, 40 mg/m2, once weekly (QW), intravenous (IV), 6 weeks and Pelvic radiation, 1.8 Gy/day, 5 days/week, 6 weeks
  Brachytherapy, 30-35 Gy over 1 week
  Interventions: Drug: Cisplatin; Radiation: Brachytherapy; Radiation: Pelvic radiation

INTERVENTIONS:
Drug: Gemcitabine
  Other Names: LY188011; Gemzar
  Arms: 1
Drug: Cisplatin
Radiation: Brachytherapy — Brachytherapy, 30-35 Gy over 1 week
Radiation: Pelvic radiation — Pelvic radiation, 1.8 Gy/day, 5 days/week, 6 weeks

SUMMARY:
The purpose of this study is to compare the effectiveness of two methods of treating cancer of the cervix. Half the patients will receive gemcitabine plus cisplatin while undergoing radiation therapy, followed by adjuvant gemcitabine and cisplatin and the other half will receive cisplatin along with radiation therapy without adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with cancer of cervix
* tumor that can be measured
* no previous treatment with chemotherapy or radiation for this cancer
* Karnofsky Performance Status Score >=70
* able to give written consent
* willing and able to participate in the study, both during the active treatment and the follow-up period.

Exclusion Criteria:

* impairment such as hearing loss from prior cisplatin therapy
* damage to nerves such as being unable to distinguish hot and cold to touch
* used other experimental medication in past 30 days
* lab test results are not within the limits required for this study
* pregnancy or breast-feeding or possibility of becoming pregnant during this study and not using an approved method of birth control.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2002-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires, Argentina
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sarajevo, Bosnia and Herzegovina
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai, India
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City, Mexico
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Karachi, Pakistan
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lima, Peru
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangkok, Thailand

REFERENCES:
- [Derived] Duenas-Gonzalez A, Zarba JJ, Patel F, Alcedo JC, Beslija S, Casanova L, Pattaranutaporn P, Hameed S, Blair JM, Barraclough H, Orlando M. Phase III, open-label, randomized study comparing concurrent gemcitabine plus cisplatin and radiation followed by adjuvant gemcitabine and cisplatin versus concurrent cisplatin and radiation in patients with stage IIB to IVA carcinoma of the cervix. J Clin Oncol. 2011 May 1;29(13):1678-85. doi: 10.1200/JCO.2009.25.9663. Epub 2011 Mar 28. PMID 21444871
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine/Cisplatin/Radiation: Gemcitabine: 125 mg/m2, once weekly (QW), intravenous (IV), 6 weeks Cisplatin: 40 mg/m2, once weekly (QW), intravenous (IV), 6 weeks Pelvic radiation: 1.8 Gy/day, 5 days/week, 6 weeks
  Brachytherapy, 30-35 Gy over 1 week
  Two week rest period with no chemotherapy or radiation
  Cisplatin, 50 mg/m2, IV, day 1 of 21 day cycle for two 21-day cycles and Gemcitabine, 1000 mg/m2, day 1 and day 8 for two 21 day cycles
- Cisplatin/Radiation: Cisplatin: 40 mg/m2, once weekly (QW), intravenous (IV), 6 weeks Pelvic radiation: 1.8 Gy/day, 5 days/week, 6 weeks
  Brachytherapy, 30-35 Gy over 1 week
Period: Overall Study
Arm/Group | Gemcitabine/Cisplatin/Radiation | Cisplatin/Radiation
Started | 259 | 256
Completed | 217 | 244
Not Completed | 42 | 12
Not completed — Adverse Event | 18 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Patient Moved | 0 | 1
Not completed — Withdrawal by Subject | 9 | 3
Not completed — Protocol Entry Criteria Not Met | 2 | 1
Not completed — Clinical Relapse | 2 | 1
Not completed — Lack of Efficacy, Progressive Disease | 1 | 2
Not completed — Lack of Efficacy, Stable Disease | 1 | 0
Not completed — Physician Decision | 3 | 1
Not completed — Death from Study Drug Toxicity | 2 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Death from Other Cause | 1 | 0
Not completed — Reason Not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine/Cisplatin/Radiation | Cisplatin/Radiation | Total
Number analyzed (Participants) | 259 | 256 | 515
Age Continuous [Mean (Standard Deviation); unit: years] | 45.8 (9.8) | 46.5 (9.2) | 46.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 256 | 515.0
  Male | 0 | 0 | 0.0
Region of Enrollment [Number; unit: participants]
  Pakistan | 27 | 29 | 56.0
  Mexico | 28 | 31 | 59.0
  Argentina | 17 | 18 | 35.0
  Thailand | 34 | 33 | 67.0
  Peru | 29 | 31 | 60.0
  India | 60 | 56 | 116.0
  Bosnia and Herzegovina | 33 | 28 | 61.0
  Panama | 31 | 30 | 61.0
Grade of Histological Diagnosis [Number; unit: participants]
  Moderately Differentiated | 114 | 119 | 233.0
  Poorly Differentiated | 48 | 44 | 92.0
  Unknown | 69 | 69 | 138.0
  Undifferentiated | 2 | 0 | 2.0
  Well Differentiated | 26 | 24 | 50.0
Karnofsky Performance Status Scale [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0-100, the lower the score, the worse the survival for most serious illnesses.
  participants
    Unknown (Missing) | 1 | 0 | 1.0
    70 - Unable to carry on normal activity | 0 | 1 | 1.0
    80 - Activity with effort; some signs of disease | 8 | 9 | 17.0
    90 - Normal activity; minor signs of disease | 147 | 145 | 292.0
    100 - Normal no complaints; no evidence of disease | 103 | 101 | 204.0
Pathological Diagnosis [Number; unit: participants]
  Adenocarcinoma of Cervix | 17 | 15 | 32.0
  Adeno/Squamous Cell Carcinoma | 198 | 199 | 397.0
  Other - Poorly Differentiated Carcinoma | 1 | 0 | 1.0
  Other - Squamous | 43 | 42 | 85.0
Race/Ethnicity [Number; unit: participants]
  Western Asian | 87 | 85 | 172.0
  Caucasian | 33 | 29 | 62.0
  East/Southeast Asian | 34 | 33 | 67.0
  Hispanic | 105 | 109 | 214.0
Stage of Disease [Number; unit: participants]
  Stage IIIA | 1 | 1 | 2.0
  Stage IIIB | 94 | 94 | 188.0
  Stage IIB | 160 | 156 | 316.0
  Stage IVA | 4 | 5 | 9.0
Height [Mean (Standard Deviation); unit: centimeters] | 155.2 (6.6) | 154.6 (6.7) | 154.9 (6.6)
Weight [Mean (Standard Deviation); unit: kilograms] | 61.2 (11.3) | 62.4 (13.0) | 61.8 (12.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progressive Disease or Death Due to Any Cause at 3 Years
Description: Original outcome was Progression-Free Survival (PFS) probability at 3 years. PFS=time from baseline to progressive disease (PD) or death from any cause. Probability is not an accepted "Measure Type", so number of progression-free patients still at risk and cumulative number of patients that had an event (PD or death of any cause) are presented.
Time Frame: Tumor assessments at baseline, weekly during chemoradiation & brachytherapy, on Day 1 of adjuvant Cycles 1&2 for Arm A, at the 30-day post-study visit, every 4/6 months for 12/48 months of the short/long post-study follow-up periods respectively
Population: Intention-to-treat population includes all randomized participants. Participants were analyzed according to treatment they were randomly assigned.
Measure: Number; unit: participants
Arm/Group | Gemcitabine/Cisplatin/Radiation | Cisplatin/Radiation
Number analyzed (Participants) | 259 | 256
participants
  3 Years: Number of Patients with Event | 55 | 83
  3 Years: Number of Patients at Risk | 149 | 141
Statistical Analysis 1: Comparison: Gemcitabine/Cisplatin/Radiation vs Cisplatin/Radiation; Test type: Superiority or Other; p = 0.029, Z Statistic — The p-value is two-sided and was tested at the 0.05 significance level; PFS Probability Difference at 3 Years = 0.095, 95% CI [0.010 to 0.179] — Difference in progression-free survival probability between Gem/Cis/Rad and Cis/Rad. The difference in PFS probability between the two treatment arms can also be presented as a percentage (ie, PFS at 3 years was 9.5% better in the Gem/Cis/Rad arm)

2. Secondary Outcome: Number of Participants With Progressive Disease or Death Due to Disease Under Study at Various Time Points
Description: Original outcome was Time to Progressive Disease (TTPD), which is the time from baseline to event (progressive disease or death due to study disease). The median TTPD was not achieved and therefore the cumulative number of participants with event (and those still at risk) at various time points are presented.
Time Frame: as for outcome 1
Population: Intent-to-treat population includes all randomized patients. Patients were analyzed according to treatment they were randomly assigned.
Measure: Number; unit: participants
Arm/Group | Gemcitabine/Cisplatin/Radiation | Cisplatin/Radiation
Number analyzed (Participants) | 259 | 256
participants
  3 Months: Number of Patients with Event | 5 | 8
  3 Months: Number of Patients at Risk | 221 | 238
  6 Months: Number of Patients with Event | 10 | 25
  6 Months: Number of Patients at Risk | 204 | 218
  12 Months: Number of Patients with Event | 21 | 44
  12 Months: Number of Patients at Risk | 186 | 195
  18 Months: Number of Patients with Event | 24 | 62
  18 Months: Number of Patients at Risk | 176 | 170
  24 Months: Number of Patients with Event | 31 | 69
  24 Months: Number of Patients at Risk | 167 | 158
  36 Months: Number of Patients with Event | 40 | 78
  36 Months: Number of Patients at Risk | 149 | 141
Statistical Analysis 1: Comparison: Gemcitabine/Cisplatin/Radiation vs Cisplatin/Radiation; Test type: Superiority or Other; p = 0.0008, Log Rank

3. Secondary Outcome: Local Failure Rate
Description: Local failure rate (LFR) was defined as the the proportion of per-protocol participants who had progressive disease (PD) in the cervix or pelvis. LFR = The number of (a) participants who progressed in the cervix or pelvis divided by (b) the number of participants in each arm. (LFR=a/b).
Time Frame: as for outcome 1
Population: Per protocol population included all randomized patients with: Histological diagnosis of cancer of cervix; No previous chemotherapy or radiation therapy; Presence of bidimensionally measurable disease, at least 2 cm in diameter; Treatment with at least one dose of study chemotherapy. Patients were analyzed according to treatment actually received.
Measure: Number; unit: proportion of participants with PD
Arm/Group | Gemcitabine/Cisplatin/Radiation | Cisplatin/Radiation
Number analyzed (Participants) | 257 | 253
proportion of participants with PD | 0.113 | 0.166
Statistical Analysis 1: Comparison: Gemcitabine/Cisplatin/Radiation vs Cisplatin/Radiation; Note: There were 2 patients with unknown site of progressive disease; these patients were counted as a Local failure. Note: There was 1 patient with both local and distant failure; this patient was counted as a Local failure; Test type: Superiority or Other; p = 0.096, Fisher Exact — The p-value is two-sided and was tested at the 0.05 significance level

4. Secondary Outcome: Tumor Response
Description: Tumor response rate (TRR) defined as number of qualified responder patients with confirmed complete or partial response.
Time Frame: as for outcome 1
Population: Qualified Responders population included all randomized patients with: Histological diagnosis of cancer of cervix; No previous chemotherapy or radiation therapy; Presence of bidimensionally measurable disease, at least 2 cm in diameter; Treatment with at least one dose of study chemotherapy. Patients were analyzed according to treatment assigned.
Measure: Number; unit: participants
Arm/Group | Gemcitabine/Cisplatin/Radiation | Cisplatin/Radiation
Number analyzed (Participants) | 256 | 254
participants
  Complete Response | 223 | 217
  Partial Response | 22 | 20
Statistical Analysis 1: Comparison: Gemcitabine/Cisplatin/Radiation vs Cisplatin/Radiation; Test type: Superiority or Other; p = 0.250, Fisher Exact — The p-value is two-sided and was tested at the 0.05 significance level

5. Secondary Outcome: Number of Participants Who Died From Any Cause at Various Time Points
Description: Original outcome was Overall Survival, which was defined as time from baseline to death from any cause.
Time Frame: baseline to date of death from any cause (includes 60 month follow-up period)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Gemcitabine/Cisplatin/Radiation | Cisplatin/Radiation
Number analyzed (Participants) | 259 | 256
participants
  3 Months: Number of Patients with Event | 3 | 0
  3 Months: Number of Patients at Risk | 253 | 254
  6 Months: Number of Patients with Event | 9 | 4
  6 Months: Number of Patients at Risk | 241 | 248
  12 Months: Number of Patients with Event | 22 | 25
  12 Months: Number of Patients at Risk | 226 | 222
  18 Months: Number of Patients with Event | 33 | 46
  18 Months: Number of Patients at Risk | 207 | 195
  24 Months: Number of Patients with Event | 39 | 58
  24 Months: Number of Patients at Risk | 200 | 182
  36 Months: Number of Patients with Event | 53 | 75
  36 Months: Number of Patients at Risk | 175 | 158
Statistical Analysis 1: Comparison: Gemcitabine/Cisplatin/Radiation vs Cisplatin/Radiation; Test type: Superiority or Other; p = 0.0224, Log Rank

6. Secondary Outcome: Number of Participants With Progressive Disease or Death Due to Any Cause at Various Time Points
Description: Original outome was Progression-Free Survival, which was defined as time from baseline to progressive disease or death due to any cause.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Gemcitabine/Cisplatin/Radiation | Cisplatin/Radiation
Number analyzed (Participants) | 259 | 256
participants
  3 Months: Number of Patients with Event | 8 | 8
  3 Months: Number of Patients at Risk | 221 | 238
  6 Months: Number of Patients with Event | 14 | 25
  6 Months: Number of Patients at Risk | 204 | 218
  12 Months: Number of Patients with Event | 29 | 45
  12 Months: Number of Patients at Risk | 186 | 195
  18 Months: Number of Patients with Event | 34 | 63
  18 Months: Number of Patients at Risk | 176 | 170
  24 Months: Number of Patients with Event | 42 | 72
  24 Months: Number of Patients at Risk | 167 | 158
  36 Months: Number of Patients with Event | 55 | 83
  36 Months: Number of Patients at Risk | 149 | 141
Statistical Analysis 1: Comparison: Gemcitabine/Cisplatin/Radiation vs Cisplatin/Radiation; Test type: Superiority or Other; p = 0.0227, Log Rank

ADVERSE EVENTS:
Arm/Group | Gemcitabine/Cisplatin/Radiation | Cisplatin/Radiation
Serious Adverse Events (participants affected / at risk) | 44 | 17
Other Adverse Events (participants affected / at risk) | 259 | 251
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Gemcitabine/Cisplatin/Radiation | Cisplatin/Radiation
Anaemia (Blood and lymphatic system disorders) | 6/260 (6) | 0/255 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 6/260 (6) | 1/255 (1)
Leukopenia (Blood and lymphatic system disorders) | 3/260 (3) | 0/255 (0)
Neutropenia (Blood and lymphatic system disorders) | 2/260 (2) | 1/255 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0/260 (0) | 1/255 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 9/260 (9) | 0/255 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1/260 (1) | 0/255 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1/260 (1) | 0/255 (0)
Blindness (Eye disorders) | 1/260 (1) | 0/255 (0)
Abdominal pain (Gastrointestinal disorders) | 4/260 (4) | 1/255 (1)
Constipation (Gastrointestinal disorders) | 0/260 (0) | 1/255 (1)
Diarrhoea (Gastrointestinal disorders) | 15/260 (17) | 3/255 (3)
Haematemesis (Gastrointestinal disorders) | 1/260 (1) | 0/255 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0/260 (0) | 1/255 (1)
Nausea (Gastrointestinal disorders) | 3/260 (3) | 3/255 (3)
Proctitis (Gastrointestinal disorders) | 4/260 (4) | 0/255 (0)
Tongue haemorrhage (Gastrointestinal disorders) | 1/260 (1) | 0/255 (0)
Vomiting (Gastrointestinal disorders) | 6/260 (6) | 4/255 (4)
Oedema (General disorders) | 1/260 (1) | 0/255 (0)
Pyrexia (General disorders) | 3/260 (3) | 2/255 (2)
Diarrhoea infectious (Infections and infestations) | 1/260 (1) | 0/255 (0)
Infection (Infections and infestations) | 1/260 (1) | 1/255 (1)
Pneumonia (Infections and infestations) | 1/260 (1) | 0/255 (0)
Sepsis (Infections and infestations) | 1/260 (1) | 0/255 (0)
Urinary tract infection (Infections and infestations) | 3/260 (3) | 3/255 (3)
Radiation skin injury (Injury, poisoning and procedural complications) | 1/260 (1) | 0/255 (0)
Blood bilirubin (Investigations) | 1/260 (1) | 0/255 (0)
Blood creatinine (Investigations) | 1/260 (1) | 0/255 (0)
Creatinine renal clearance decreased (Investigations) | 2/260 (2) | 0/255 (0)
Dehydration (Metabolism and nutrition disorders) | 2/260 (2) | 1/255 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0/260 (0) | 1/255 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 6/260 (7) | 1/255 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1/260 (1) | 0/255 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 5/260 (5) | 1/255 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1/260 (1) | 0/255 (0)
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/260 (1) | 0/255 (0)
Cerebral ischaemia (Nervous system disorders) | 0/260 (0) | 1/255 (1)
Depressed level of consciousness (Nervous system disorders) | 0/260 (0) | 1/255 (1)
Leukoencephalopathy (Nervous system disorders) | 1/260 (1) | 0/255 (0)
Dysuria (Renal and urinary disorders) | 0/260 (0) | 1/255 (1)
Haematuria (Renal and urinary disorders) | 1/260 (1) | 0/255 (0)
Renal failure (Renal and urinary disorders) | 1/260 (1) | 1/255 (1)
Renal failure acute (Renal and urinary disorders) | 0/260 (0) | 1/255 (1)
Urethral obstruction (Renal and urinary disorders) | 1/260 (1) | 0/255 (0)
Pelvic pain (Reproductive system and breast disorders) | 0/260 (0) | 1/255 (1)
Vaginal fistula (Reproductive system and breast disorders) | 1/260 (1) | 0/255 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 5/260 (5) | 5/255 (5)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0/260 (0) | 1/255 (1)
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1/260 (1) | 0/255 (0)
Deep vein thrombosis (Vascular disorders) | 2/260 (2) | 0/255 (0)
Hypertension (Vascular disorders) | 1/260 (1) | 0/255 (0)
Hypotension (Vascular disorders) | 0/260 (0) | 1/255 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Gemcitabine/Cisplatin/Radiation | Cisplatin/Radiation
Anaemia (Blood and lymphatic system disorders) | 175/260 (233) | 115/255 (130)
Leukopenia (Blood and lymphatic system disorders) | 145/260 (271) | 114/255 (124)
Lymphopenia (Blood and lymphatic system disorders) | 31/260 (41) | 31/255 (32)
Neutropenia (Blood and lymphatic system disorders) | 193/260 (378) | 74/255 (78)
Thrombocytopenia (Blood and lymphatic system disorders) | 66/260 (79) | 30/255 (30)
Abdominal pain (Gastrointestinal disorders) | 87/260 (115) | 57/255 (64)
Constipation (Gastrointestinal disorders) | 44/260 (47) | 34/255 (36)
Diarrhoea (Gastrointestinal disorders) | 159/260 (207) | 131/255 (151)
Dyspepsia (Gastrointestinal disorders) | 19/260 (19) | 14/255 (17)
Nausea (Gastrointestinal disorders) | 167/260 (280) | 155/255 (179)
Proctalgia (Gastrointestinal disorders) | 20/260 (22) | 16/255 (16)
Proctitis (Gastrointestinal disorders) | 47/260 (52) | 25/255 (25)
Vomiting (Gastrointestinal disorders) | 146/260 (248) | 121/255 (138)
Asthenia (General disorders) | 28/260 (37) | 9/255 (9)
Fatigue (General disorders) | 80/260 (126) | 57/255 (67)
Pyrexia (General disorders) | 31/260 (38) | 21/255 (21)
Cystitis (Infections and infestations) | 17/260 (19) | 10/255 (10)
Vaginal infection (Infections and infestations) | 29/260 (33) | 22/255 (25)
Radiation skin injury (Injury, poisoning and procedural complications) | 72/260 (77) | 65/255 (67)
Alanine aminotransferase (Investigations) | 19/260 (23) | 7/255 (8)
Aspartate aminotransferase (Investigations) | 22/260 (26) | 4/255 (4)
Creatinine renal clearance decreased (Investigations) | 62/260 (81) | 51/255 (59)
Anorexia (Metabolism and nutrition disorders) | 53/260 (61) | 44/255 (46)
Back pain (Musculoskeletal and connective tissue disorders) | 29/260 (34) | 30/255 (32)
Myalgia (Musculoskeletal and connective tissue disorders) | 16/260 (18) | 8/255 (9)
Headache (Nervous system disorders) | 38/260 (47) | 23/255 (25)
Dysuria (Renal and urinary disorders) | 95/260 (114) | 80/255 (85)
Pollakiuria (Renal and urinary disorders) | 17/260 (17) | 14/255 (15)
Genital discharge (Reproductive system and breast disorders) | 20/260 (21) | 17/255 (17)
Pelvic pain (Reproductive system and breast disorders) | 71/260 (80) | 63/255 (68)
Vaginal discharge (Reproductive system and breast disorders) | 70/260 (84) | 62/255 (62)
Vaginal haemorrhage (Reproductive system and breast disorders) | 148/260 (157) | 157/255 (162)
Cough (Respiratory, thoracic and mediastinal disorders) | 18/260 (18) | 15/255 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 14/260 (16) | 9/255 (9)
Hypertension (Vascular disorders) | 19/260 (19) | 21/255 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days